CLINICAL TRIAL: NCT07031089
Title: City-hospital Collaboration for the Early Screening of Hepatic Fibrosis in Primary Care: a Secondary Prevention Project in the Grenoble Health Basin
Acronym: PREFIB
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A010187-42
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional study (RIPH category 3) — The study aims to describe and evaluate an existing care pathway, implemented within the framework of current clinical practice, without modifying the modalities of care or adding specific interventions. No additional procedures are imposed on participants, apart from data collection for evaluation purposes and telephone interviews.

SUMMARY:
Cirrhosis and hepatocellular carcinoma (HCC) are responsible for 25,000 deaths per year in France. The main causes are excessive alcohol consumption, metabolic steatosis, and hepatitis B and C. Fibrosis, classified from F0 (absence of fibrosis) to F4 (cirrhosis), is the sole determinant of liver-related mortality, particularly from stage F3. The incidence of metabolic steatosis is increasing, associated with a rise in mortality from chronic liver diseases (CLD). CLDs, often asymptomatic, are diagnosed late, reducing patient survival. Recommendations exist for the screening of hepatic fibrosis in at-risk patients (alcohol, diabetes, metabolic syndrome). This screening relies on calculating the FIB-4 score (calculated from widely prescribed variables: AST, ALT, platelets, age), followed by Fibroscan® (a non-invasive test for hepatic fibrosis) if FIB-4 > 1.3.

A Fibroscan® result <8kPa excludes advanced fibrosis, while a result >9.6kPa suggests advanced fibrosis and ≥15kPa indicates cirrhosis. The appropriate care pathway includes a risk reduction program, a specialized consultation for patients with Fibroscan® ≥8kPa, and semi-annual screening for HCC in the case of cirrhosis. Indeed, it has been shown in a French cohort of patients with viral C cirrhosis that adherence to semi-annual screening is associated with better survival.

Eligible patients are primarily seen in primary care, and INCA has published a recommendation intended for general practitioners to improve the screening of fibrosis [13]. However, FIB-4 is poorly known among general practitioners [14], and access to Fibroscan® remains limited [15], hindering the implementation of the recommendations. Therefore, a care pathway has been established in the Grenoble area, initiated by Professor Costentin, allowing access to Fibroscan® for patients in primary care, starting from 2022 at the CHU. The objective is to evaluate the completion of the pathway, particularly the management of MCF risk factors and referral to specialized consultation for patients with Fibroscan® ≥8 kPa.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Having undergone a Fibroscan® at the CHU de Grenoble-Alpes , requested by a primary care practitioner (general practitioner, non-hospital diabetologist, Asalée nurse), as part of the screening recommendations for liver fibrosis in the case of a FIB4 score > 1.3
* With a result ≥ 8kPa
* Between January 2023 and January 2026

Exclusion Criteria:

* Patients who have expressed their opposition to participating in the study
* Patients under guardianship or deprived of liberty
* Patients with a known chronic liver disease who are being monitored at the time of the Fibroscan® procedure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the Grenoble area underwent a Fibroscan® at CHU Grenoble Alpes, upon request by a primary care practitioner, as part of hepatic fibrosis screening (FIB-4 >1.3, Fibroscan® ≥8kPa). Eligible patients will be contacted by a clinical research associate for a telephone questionnaire, with the possibility of questioning the prescribing physician.
  Between January 2023 and January 2025, 264 patients were referred: 178 to CHU Results:
  30% Fibroscan® ≥8kPa (eligible for specialized consultation)
  18% Fibroscan® >9.6kPa (probable advanced fibrosis F3F4)
  10% Fibroscan® ≥15kPa (probable cirrhosis)
  Projections: 500 patients will undergo Fibroscan® between 2023 and 2026, with 150 having a result ≥8kPa.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-11-02 (Estimated); Primary Completion 2028-05-02 (Estimated); Study Completion 2028-11-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of managment of risk factors for significant liver fibrosis. | Up to 30 months
  Proportion of patients with Fibroscan® ≥ 8kPa who received a specialized consultation in hepatogastroenterology in the year following the Fibroscan®

SECONDARY OUTCOMES:
Frequency of risk factors for liver fibrosis. | Up to 30 months
  proprtion of patient with risk factors for liver fibrosis.
Evaluation of managment of risk factors for liver fibrosis. | Up to 30 months
  Proportion of patients who received appropriate management of identified risk factors.
Evaluation of patients satisfaction after | Up to 30 months
  Proportion of patients who satisfied with their care pathway evaluted with the 'patient' satisfaction and difficulties questionnaire .
Evaluation of social determinals of health associated to the risks of advanced of liver fibrosis. | up to 30 months
  Estimation of the risks of advanced liver fibrosis according to the above definition associated with predefined variables of interest.
Evaluation of managment of risk factors for significant liver fibrosis in chu Grenoble Alpes patients . | up to 30 months
  Main judgment criterion estimated among patients screened at the university hospital.
Evaluation of the proportion of patients who had at least one specialized consultation within 12 months. | up to 30 months
  Proportion of patients who had at least one specialized consultation in 12 months.